CLINICAL TRIAL: NCT00484679
Title: Adrenal Function and Use of Intralesional Triamcinolone Acetonide 10 mg/mL (Kenalog-10) in Patients With Alopecia Areata
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Alopecia Areata Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 0609M91989
Record Dates: First submitted 2007-06-08; First posted 2007-06-11 (Estimated); Results first posted 2014-06-20 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2017-04

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — Triamcinolone Acetonide; Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients receiving Triamcinolone Acetonide 10 ml (Kenalog-10) intralesional injections.
  Interventions: Drug: Triamcinolone Acetonide 10 mg/mL (Kenalog-10)

INTERVENTIONS:
Drug: Triamcinolone Acetonide 10 mg/mL (Kenalog-10) — Triamcinolone Acetonide 10 mg/ml (Kenalog-10) intralesional injection
  Other Names: Kenalog 10

SUMMARY:
The purpose of the study is to see whether treating alopecia areata with injections of the corticosteroid, Triamcinolone acetonide 10mg/cc (Kenalog-10), has an impact on the adrenal glands.

DETAILED DESCRIPTION:
1. To determine the effects of intralesional Triamcinolone Acetonide 10mg/cc (Kenalog 10) use for the treatment of alopecia areata on adrenal function.
2. To evaluate the efficacy of intralesional corticosteroids (Kenalog-10)on hair regrowth in moderate to severe alopecia areata.

18 subjects with moderate to severe alopecia areata were enrolled and 15 subjects completed all study visits.

Subjects underwent intralesional triamcinolone acetonide (10mg/cc) (Kenalog-10) injections every 6 weeks for a period of 6 months in the General Clinical Research Center (GCRC). This period was followed by a 6 week, injection-free, safety follow-up visit. Adrenal function was assessed by utilization of the Low Dose Adrenocorticotropic Hormone Stimulation Test (ACTH) which measures adrenal gland production of cortisol after exogenously administered ACTH. Serum blood draws of 3 mL were done at baseline and 6-week intervals at the start of each scheduled appointment for intralesional treatment at approximately 0800 hours. Two blood draws were taken at time 0 and again 30 minutes after a 1 mcg bolus dose of synthetic ACTH (Cortrosyn).

Patients underwent their scheduled course of intralesional corticosteroid (Kenalog-10) injections and other study data was collected, such as SALT scores and physician assessments of AA, during the time between blood draws.

ELIGIBILITY:
Inclusion Criteria:

* Subject has clinical diagnosis of alopecia areata.
* Written informed consent and HIPAA authorization have been obtained.

  * Female subjects of childbearing potential have a negative pregnancy test and agree to use an acceptable method of birth control to prevent pregnancy.
* In the opinion of the investigator, subject is a candidate for intralesional therapy for alopecia areata.
* Subject agrees to comply with protocol requirements and attend all required study visits and is considered to be a good study subject.
* Subject meets concomitant medication washout requirements.
* Subject is >/= 18 years of age.

Exclusion Criteria:

* Subject has alopecia universalis.
* Subject has known adrenocortical insufficiency or Cushing's Syndrome.
* Subject is pregnant or lactating.
* Subject has current controlled or uncontrolled bacterial, viral, fungal, atypical, or opportunistic infections.
* Subject possesses hypersensitivity to cortrosyn or Triamcinolone Acetonide (Kenalog-10) or any component of their formulation.
* Subject is currently or has undergone therapy for malignancy within the past five years.
* Subject has history of substance abuse within the past five years.
* Subject has used oral corticosteroids within the past 12 months.
* Subject has concurrent use of phenytion rifampin, phenobarbital, mitotane, or other formulations of corticosteroid medications.
* Subject has any medical condition that, in the judgement of the investigator, would jeopardize the subject's safety following exposure to the administered medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-05; Primary Completion 2009-06 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria K Hordinsky, MD, Study Director — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- (Kenalog-10) Intralesional Injections for Alopecia Areata: Patients received Triamcinolone Acetonide 10 ml (Kenalog-10) intralesional injections every 6 weeks for 6 months. Disease extent and efficacy was assessed along with safety studies involving regularly scheduled ACTH stimulation tests.
Period: Overall Study
Arm/Group | (Kenalog-10) Intralesional Injections for Alopecia Areata
Started | 18
Completed | 15
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: 15 completed the study and were used for analysis.
Arm/Group | (Kenalog-10) Intralesional Injections for Alopecia Areata
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (14.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Cortisol Levels From Baseline to Week 24
Description: Mean change in cortisol levels from baseline to week 24 after four triamcinolone acetonide 10 ml injections 6 weeks apart.
Time Frame: baseline, week 24
Population: Participants who completed all treatment and follow-up visits
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | (Kenalog-10) Intralesional Injections for Alopecia Areata
Number analyzed (Participants) | 15
mg/dL | 0.187 (6.019)

ADVERSE EVENTS:
Arm/Group | (Kenalog-10) Intralesional Injections for Alopecia Areata
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 17/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | (Kenalog-10) Intralesional Injections for Alopecia Areata (N=18)
acne (Skin and subcutaneous tissue disorders) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1)
atrophy of scalp (Skin and subcutaneous tissue disorders) | 2 (2)
benign keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Broken left elbow (Musculoskeletal and connective tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
erythema of ear canal (Ear and labyrinth disorders) | 2 (2)
excoriations (Skin and subcutaneous tissue disorders) | 2 (2)
facial flushing (Skin and subcutaneous tissue disorders) | 2 (3)
feelings of sadness (Psychiatric disorders) | 1 (3)
influenza (Infections and infestations) | 1 (1)
folliculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Headaches (General disorders) | 4 (6)
increased number of telantascias along frontal hair line (Skin and subcutaneous tissue disorders) | 1 (1)
Increase scalp hair loss (Skin and subcutaneous tissue disorders) | 1 (1)
Irregular periods (Reproductive system and breast disorders) | 2 (2)
conjunctivitis (Eye disorders) | 1 (1)
throat erythema (Respiratory, thoracic and mediastinal disorders) | 2 (3)
nasal septal fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
intermittant nose bleeds (General disorders) | 1 (1)
pinguecula (Eye disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Restless leg syndrome (Nervous system disorders) | 1 (1)
scale in ear canal (Skin and subcutaneous tissue disorders) | 1 (1)
tonsilar gland enlargement (General disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 (3)
vaginal bleeding (Reproductive system and breast disorders) | 2 (2)
vaginal yeast infection (Infections and infestations) | 1 (1)
worsening ear dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
xerotic skin (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No